CLINICAL TRIAL: NCT06671691
Title: Phase I Dose-Escalation Clinical Trial of Definitive Single Dose Stereotactic Body Radiotherapy in Patients with Low-risk Hormone Receptor-positive and Her2-negative Breast Cancer Not Suitable or Who Refuse Surgery: DESERT I Trial
Brief Title: A Phase I Dose-escalation Trial of Definitive Single Dose Stereotactic Body Radiotherapy in Low-risk Breast Cancer Patients: DESERT I Trial
Acronym: DESERT-I
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Universitat de les Illes Balears (Other)
Responsible Party: Principal Investigator, Jon Gadea Quinteiro, Radiation Oncologist, Universitat de les Illes Balears
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IB 5560/24 PI
Record Dates: First submitted 2024-10-28; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3); SBRT
Keywords: Breast cancer; SBRT; Radiotherapy; early stage; Definitive treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Treatment tolerance will be the basis for allowing us to progress to the next dose level.
  Dose-limiting toxicity (DLT) will be defined as a G3-G4 toxicity or G2 in cases of hypo/hyperpigmentation according to the CTCAE v5.0 scale, assessing the following items: induration, ulceration, pruritus, pigmentation changes, and fatigue. If, at 3 months post-RT at the initial dose level, none of the patients present a DLT, three new patients will receive RT at the next dose level. However, if any patient in a group presents a DLT, three additional patients will be added at the same dose level. Dose escalation will continue up to 30Gy unless >33% of patients in a single dose group experience a DLT.
  If >33% of patients at a dose level experience a DLT, the study will end, and the dose level immediately below this will be selected to design the phase II of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- SBRT level I: 20Gy (Experimental): 20Gy in 1 fraction will be delivered to the tumor
  Interventions: Radiation: SBRT level I
- SBRT level II: 23Gy (Experimental): 23Gy in 1 fraction will be delivered to the tumor
  Interventions: Radiation: SBRT level II
- SBRT level III: 26Gy (Experimental): 26Gy in 1 fraction will be delivered to the tumor
  Interventions: Radiation: SBRT level III
- SBRT level IV: 28Gy (Experimental): 28Gy in 1 fraction will be delivered to the tumor
  Interventions: Radiation: SBRT level IV
- SBRT level V: 30Gy (Experimental): 30Gy in 1 fraction will be delivered to the tumor
  Interventions: Radiation: SBRT level V

INTERVENTIONS:
Radiation: SBRT level I — 20Gy in 1 fraction will be tested on the tumor using stereotactic body radiotherapy (SBRT) technique
  Arms: SBRT level I: 20Gy
Radiation: SBRT level II — 23Gy in 1 fraction will be tested on the tumor using stereotactic body radiotherapy (SBRT) technique
  Arms: SBRT level II: 23Gy
Radiation: SBRT level III — 26Gy in 1 fraction will be tested on the tumor using stereotactic body radiotherapy (SBRT) technique
  Arms: SBRT level III: 26Gy
Radiation: SBRT level IV — 28Gy in 1 fraction will be tested on the tumor using stereotactic body radiotherapy (SBRT) technique
  Arms: SBRT level IV: 28Gy
Radiation: SBRT level V — 30Gy in 1 fraction will be tested on the tumor using stereotactic body radiotherapy (SBRT) technique
  Arms: SBRT level V: 30Gy

SUMMARY:
Radiotherapy (RT) is a fundamental pillar in the fight against cancer. In the case of breast cancer, RT has traditionally been applied as an adjuvant treatment following surgery. However, in recent years, there has been research into the potential benefit of administering RT prior to surgery in a neoadjuvant manner. Given that these studies have shown promising results, it is logical to think that certain patients could benefit from exclusive RT treatment, thereby avoiding surgery and its possible sequelae. This study is a phase I dose-escalation clinical trial with sequential assignment, open-label, in which five different doses (20Gy, 23Gy, 26Gy, 28Gy, and 30Gy) will be tested on the tumor using stereotactic body radiotherapy (SBRT) technique.

The aim of the study is to determine the maximum tolerated dose (MTD) based on acute toxicity, which will allow us to proceed with a phase II clinical trial to confirm efficacy and assess the late toxicity of the treatment. Secondary objectives include assessing the pathological response via core needle biopsy (CNB), radiological response, quality of life, and cosmesis. Additionally, molecular studies will be conducted on tissue and through liquid biopsy; pre- and post-treatment, we aim to identify mutations and predictors of response.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Female gender
* ECOG score 0-2
* Positive biopsy for invasive non-lobular breast tumor histology
* Tumor < 3 cm in diameter as measured by MRI or contrast mammography
* Tumor located ≥ 0.5 cm from the skin or rib cage, clinically or radiologically
* Positive estrogen and/or progesterone receptors
* HER2 negative
* No lymphovascular invasion in the biopsy
* Tumor must be clinically and radiologically N0 (no lymph node involvement). If a suspicious lymph node is seen, it must be biopsied and show a negative result
* Patient weight below 220 kg (weight limit for the treatment table)
* Ability to tolerate the supine position for 20 minutes during treatment
* Able to undergo MRI and/or contrast mammography
* Not pregnant; women of childbearing potential will undergo a pregnancy test to rule this out
* Contraindication to or refusal of surgical treatment, which must be explicitly documented in the medical record.

Exclusion Criteria:

* Under 18 years of age
* Male gender
* ECOG score 3-4
* Positive biopsy for invasive lobular carcinoma or ductal carcinoma in situ
* Tumor ≥ 3 cm in diameter as measured by MRI
* Tumor located < 0.5 cm from the skin or rib cage, clinically or radiologically
* Negative estrogen and progesterone receptors
* HER2 positive
* Presence of lymphovascular invasion in the biopsy
* Positive BRCA mutation
* Multicentric tumor
* Tumor with positive axillary lymph nodes
* Patients with metastatic disease
* History of previous breast cancer in the same breast
* Previous thoracic radiotherapy
* Pregnant or actively breastfeeding
* Unable to undergo MRI or contrast mammography
* Unable to tolerate the supine position
* Patient with breast implants
* Patients with pacemakers
* Scleroderma, lupus, or other connective tissue diseases with active flares
* Inability to understand and sign the informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Establish the single-fraction radiation dose (MTD) | 3 months
  To establish the single-fraction SBRT radiation dose (MTD) that causes an incidence of dose-limiting toxicities (DLTs) lower than 33%

SECONDARY OUTCOMES:
Chronic toxicity | 1 year
  Assessed at 6 and 12 months post-treatment using CTCAE v5.0 criteria for skin, fatigue, and breast.
Radiological response to treatment | 1 year
  Measured with MRI or contrast mammography 12 months post-RT using RECIST criteria.
Pathological response to treatment | 1 year
  Between 1 and 3 core needle biopsies (CNB) will be performed, guided by ultrasound on the treated lesion at 6 and 12 months post-RT to establish the rate of residual tumor cells scored by pathology review of H&E slides.
Patient-reported quality of life | 1 year
  Measured using the EORTC QLQ-C30 questionnaires before RT and at 3 and 12 months post-treatment.
  EORTC QLQ-C30- scale goes from 1/not at all to 4/very much. There is additionally a rate of overall health and quality of life that is a scale from 1 to 7.
Cosmesis after treatment | 1 year
  Measured using the Modified Harvard-Harris Cosmetic Scale (MHHCS) at 1, 3, 6, and 12 months post-treatment. Photographs of the breasts will be taken before treatment and at each follow-up visit, to be evaluated later using an external validation system.
  The MHCCS scale compares baseline images with those obtained post-treatment, allowing the assessment of cosmesis as follows: Poor, fair, good or excellent.
Tumor DNA sequencing | 1 year
  Tumor biopsies will be taken before and at 6 and 12 months post-treatment. Next Generation Sequencing (NGS) will be performed to characterize radiation-induced changes in tumor DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Gadea Quinteiro, Principal investigator, Principal Investigator — Universitat de les Illes Balears
Locations (1):
- Hospital Universitario Son Espases, Palma, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No